CLINICAL TRIAL: NCT01023815
Title: Once-a-day Regimen or Steroid Withdrawal in de Novo Kidney Transplant Recipients Treated With Everolimus, Cyclosporine and Steroids: a 12-month, Prospective, Randomized, Multicenter, Open-label Study. The EVIDENCE Study (EVerolImus Once-a-Day rEgimen With Neoral Versus Corticosteroid Elimination).
Brief Title: Once-a-day Regimen With Everolimus, Low Dose Cyclosporine and Steroids in Comparison With Steroid Withdrawal or Twice a Day Regimen With Everolimus, Low Dose Cyclosporine and Steroids.
Acronym: EVIDENCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001AIT12
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Results first posted 2013-11-14 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-06

CONDITIONS: de Novo Kidney Transplant Recipients; Renal Transplantation
Keywords: Immunosuppression; renal transplantation; once-a-day regimen; steroid withdrawal; drug minimization; immunosuppression for prevention of acute rejections
MeSH Terms: interventions — Everolimus; Cyclosporine

ARMS (4):
- Group A -Once-a-day regimen (Experimental): Everolimus: in patients randomized to Group A before Amendment 1 approval, from the day following randomization, the whole daily dose of everolimus was taken in the morning, at the same time of the CsA and steroid dosing. At the Rand+1W visit, the everolimus dose was adjusted to reach and maintain everolimus blood levels between 5 and 8 ng/mL until end of Month 12.
  Cyclosporine: in patients randomized to Group A before Amendment 1 approval, from the day following randomization, the whole cyclosporine daily dose was taken in the morning. The dose was then adjusted to maintain C2 levels between 350 and 700 ng/mL.
  Prednisone: In patients randomized to Group A before Amendment 1 approval, the dose of prednisone was kept stable at 5 mg/day in the morning.
  Interventions: Drug: everolimus; Drug: cyclosporine; Drug: Prednison (continuous steroids)
- Group B - Steroid Withdrawal group (Experimental): Everolimus: after randomization the everolimus dose was adjusted, if necessary, to maintain a C0 within 6-10 ng/mL until M12.
  Cyclosporine:after randomization the cyclosporine dose was adjusted to maintain CsA C2 levels within 300-500 ng/mL until M12.
  Prednisone: starting from Visit 5 (day 90 ± 28 days), oral prednisone was tapered until complete stop. It was recommended to taper prednisone by 1 mg/week until complete stop in 5 to 6 weeks.
  Interventions: Drug: everolimus; Drug: cyclosporine; Drug: Prednison (continuous steroids)
- Group C - Standard twice-a-day group (Active Comparator): Everolimus: after randomization the everolimus dose was adjusted, if necessary, in order to maintain a C0 within 6-10 ng/mL until M12.
  Cyclosporine: after randomization the cyclosporine dose was gradually adjusted to reach and maintain C2 blood levels of 200-450 ng/mL between Month 6 and Month 12.
  Prednisone: the dose of prednisone was kept stable at 5 mg/day in the morning.
  Interventions: Drug: everolimus; Drug: cyclosporine; Drug: Prednison (continuous steroids)
- Not Randomized Population (NRP) (Experimental): NRP defined in whom a renal transplantation was performed, received at least one dose of study drug (everolimus) but who did not qualify for randomization at Visit 5, Day 90. This group was addressed as "not randomized patients" (NRP) and described with respect to baseline characteristics, treatment and outcome variables.
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus — Everolimus (Certican®) was provided in blisters containing tablets of 0.25 mg and 0.75 mg. Everolimus was initiated within 48 hours after graft reperfusion and it was administered orally.
  Other Names: Certican®)
Drug: cyclosporine — Cyclosporine for microemulsion (CsA, Sandimmun® Neoral®) was coadministered with everolimus at the same time of the day. CsA was available in alu-alu blisters containing soft gelatine capsules of 100 mg, 50 mg, 25 mg and 10 mg. Oral solution, as bottles containing 50 mL of solution (100 mg/mL) has been provided and used in case the drug had been administered to patients by nasogastric tube immediately after transplant.
  Other Names: CsA, Sandimmun® Neoral®
  Arms: Group A -Once-a-day regimen; Group B - Steroid Withdrawal group; Group C - Standard twice-a-day group
Drug: Prednison (continuous steroids) — continuous steroids
  Arms: Group A -Once-a-day regimen; Group B - Steroid Withdrawal group; Group C - Standard twice-a-day group

SUMMARY:
This study will compare the following immunosuppressive regimens in recipients of kidney transplantation: A) everolimus, cyclosporine and steroids given once-a-day; B) everolimus and cyclosporine given twice a day with steroid withdrawal; C) everolimus, cyclosporine given twice a day and continuous steroids. The purpose of this study is to evaluate regimens A and B in comparison with the control group (group C) for efficacy, using as main endpoint the treatment failure rate, a composite endpoint including death, graft loss, BPAR and lost to follow-up between randomization and Month 12.

ELIGIBILITY:
Inclusion criteria:

* recipients of 1st or 2nd single kidney transplant
* donor age >14 years
* females capable of becoming pregnant must have a negative serum pregnancy test within 7 days prior to or at Baseline (Visit 2), and are required to practice an approved method of birth control for the duration of the study and for a period of 2 months following discontinuation of study medication
* patientswho are willing and able to participate in the study and from whom written informed consent has been obtained

Exclusion criteria:

Exclusion criteria at screening (pre-transplantation, Visit 1):

* recipients of kidney-pancreas transplant, double kidney or any other transplant
* recipients of a 2nd kidney transplant who lost the 1st for immunological reasons
* focal segmental glomerulosclerosis (FSGS), primary oxaluria or other diseases (as cause of end stage renal failure - ESRF) at high risk of rapid recurrence or requiring continuous corticosteroid treatment
* recipients of A-B-O incompatible transplants
* historical or current peak PRA of >25% (current = 3 months)
* patients with already existing antibodies against the donor
* thrombocytopenia (platelets <75,000/mm³), absolute neutrophil count of <1,500/mm³, leucopenia (leucocytes <2,500/mm³), or hemoglobin <6 g/dL
* symptoms of significant somatic or mental illness. Inability to cooperate or communicate with the investigator, or to comply with the study requirements, or to give informed consent
* history of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases
* patients who are HIV positive or Hepatitis B surface antigen positive (HbsAg); HCV positive patients receiving interferon and/or ribavirin
* evidence of severe liver disease (incl. abnormal liver enzyme profile, i.e. AST, ALT or total bilirubin >3 times UNL)
* evidence of drug or alcohol abuse
* body mass index (BMI) >35
* patients who need to be treated with drugs known to strongly interact with CsA and/or everolimus (as detailed in Appendix 2 of the protocol) should be excluded, if according the investigator this interferes with the objectives of the study
* women of child-bearing potential, UNLESS they are using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method
* pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>5 mIU/mL)
* use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
* history of hypersensitivity to any of the study drugs or to drugs of similar chemical classes
* patients with severe active infections or any other medical condition(s) that in the view of the investigator prohibits participation in the study (specify as required)

Additional exclusion criteria post-transplantation (Visit 2):

• graft not perfused or with thrombosis of the main vessels, according to angioscintigraphy or echocolordoppler within 48 hours after the end of surgical procedure

To avoid any possible influence of the confounding factors on the results of this study additional exclusion criteria at randomization were (Visit 5, Month 3):

* unsatisfactory renal function (CrCl according Cockcroft and Gault<40 mL/min)
* proteinuria ≥0.8 g/24 hrs
* steroid-resistant, humoral, moderate/severe (BANFF grade ≥II) biopsy proven acute rejections
* multiple (2 or more) biopsy proven or treated acute rejections or acute rejections leading to relevant loss of renal function
* acute rejection or impairment of renal function (increase of serum creatinine>30%) in the month preceding randomization
* severe/uncontrollable adverse events with suspected relationship to everolimus (e.g. anemia, oral aphtosis, arthralgia) for the control of which the investigator has planned the withdrawal of everolimus
* severe infections requiring hospitalization in the two weeks preceding randomization
* poor compliance to prescribed treatments

  * Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2009-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- Italy (28):
  - Novartis Investigative Site, Perugia, Perugia
  - Novartis Investigative Site, Sassari, Sassari
  - Novartis Investigative Site, Ancona
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Brescia
  - Novartis Investigative Site, Cagliari
  - Novartis Investigative Site, Catania
  - Novartis Investigative Site, Coppito
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Modena
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Novara
  - Novartis Investigative Site, Padua
  - Novartis Investigative Site, Palermo
  - Novartis Investigative Site, Parma
  - Novarits Investigative Site, Pisa
  - Novartis Investigative Site, Roma
  - Novartis Investigative Site, Rome
  - Novartis Investigative Site, Salerno
  - Novartis Investigative Site, Siena
  - Novartis Investigative Site, Torino
  - Novartis Investigative Site, Treviso
  - Novartis InvestigativeSite, Udine
  - Novartis Investigative Site, Varese
  - Novartis Investigative Site, Verona
  - Novartis Investigative Site, Vicenza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 332 patients were screened. 330 were pre-randomized, 2 were not. Additionally, 2 pts were not treated which made the safety/ITT population 328. Of the 328, 184 were randomized and 144 were not. Of the 144, 70 dropped before day 90 & 74 completed the pre-rand period but were not randomized because they were not eligible for randomization.
Pre-assignment Details: During the Pre-randomization Period all patients received the same treatments. At V5 eligible patients were randomized 1:1:1 to one of the treatment arms and entered the Randomized Treatment Period. After Amendment 1 approval, randomization to once-a-day regimen group was stopped and patients were randomized 1:1 to Group B or Group C.
Groups:
- Pre-randomized: Not-randomization Patients (NRP): At the Baseline visit, performed up to 48 hours after graft reperfusion, eligible patients entered the Pre-Randomization Period and started study drug treatment (D1 = 1st day of everolimus treatment).
  Not-randomization Patients (NRP) was defined in whom a renal transplantation was performed, received at least one dose of study drug (everolimus) but who did not qualify for randomization at Visit 5, Day 90. This group was addressed as "not randomized patients" (NRP)
- Randomized: Group A - Once-a-day Regimen: Change in study design (Amendment 1) stopped the randomization into Group A (once-a-day regimen), due to overall slow enrollment rate and shifted all relative objectives from primary/secondary to exploratory, due to small sample size.
  Everolimus: in patients randomized to Group A before Amend 1 approval, from the day following randomization, the whole daily dose of everolimus was taken in the morning, at the same time of the CsA and steroid dosing. At the Rand+1W visit, the everolimus dose was adjusted to reach and maintain everolimus blood levels between 5 and 8 ng/mL until end of Month 12.
  Cyclosporine: in patients randomized to Group A before Amend 1 approval, from the day following randomization, the whole cyclosporine daily dose was taken in the morning. The dose was then adjusted to maintain C2 levels between 350 and 700 ng/mL.
  Prednisone: In patients randomized to Group A before Amend 1 approval, the dose of prednisone was kept stable at 5 mg/day in the morning.
- Randomized: Group B - Steroid Withdrawal Group: Everolimus: after randomization the everolimus dose was adjusted, if necessary, to maintain a C0 within 6-10 ng/mL until M12.
  Cyclosporine: after randomization the cyclosporine dose was adjusted to maintain CsA C2 levels within 300-500 ng/mL until M12.
  Prednisone: starting from Visit 5 (day 90 ± 28 days), oral prednisone was tapered until complete stop. It was recommended to taper prednisone by 1 mg/week until complete stop in 5 to 6 weeks.
- Randomized: Group C - Standard Twice-a-day Group: Everolimus: after randomization the everolimus dose was adjusted, if necessary, in order to maintain a C0 within 6-10 ng/mL until M12.
  Cyclosporine: after randomization the cyclosporine dose was gradually adjusted to reach and maintain C2 blood levels of 200-450 ng/mL between Month 6 and Month 12.
  Prednisone: the dose of prednisone was kept stable at 5 mg/day in the morning.
Period: Pre-randomization Period (Day 1 to 90)
Arm/Group | Pre-randomized: Not-randomization Patients (NRP) | Randomized: Group A - Once-a-day Regimen | Randomized: Group B - Steroid Withdrawal Group | Randomized: Group C - Standard Twice-a-day Group
Started | 328 (Out of 330 enrolled, 2 patients never received everolimus.) | 0 | 0 | 0
Completed | 184 | 0 | 0 | 0
Not Completed | 144 | 0 | 0 | 0
Not completed — Did not meet inclusion criteria | 144 | 0 | 0 | 0
Period: Randomized Period (Day 90 to Month 12)
Arm/Group | Pre-randomized: Not-randomization Patients (NRP) | Randomized: Group A - Once-a-day Regimen | Randomized: Group B - Steroid Withdrawal Group | Randomized: Group C - Standard Twice-a-day Group
Started | 0 | 45 (Randomized patients to Group A, B and C are also intent to treat population.) | 68 | 71
Completed | 0 | 42 | 60 | 68
Not Completed | 0 | 3 | 8 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Administrative Problems | 0 | 1 | 6 | 2
Not completed — Graft Loss | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: The Safety Population (SAF population) includes all patients who signed an informed consent, performed renal transplantation and received at least one dose of study drug (everolimus).
Groups:
- Not Randomized Population (NRP): At the Baseline visit, performed up to 48 hours after graft reperfusion, eligible patients entered the Pre-Randomization Period and started study drug treatment (D1 = 1st day of everolimus treatment).
  Not-randomization Patients (NRP) was defined in whom a renal transplantation was performed, received at least one dose of study drug (everolimus) but who did not qualify for randomization at Visit 5, Day 90. This group was addressed as "not randomized patients" (NRP)
- Group A - Once-a-day Regimen: Change in study design (Amendment 1) stopped the randomization into Group A (once-a-day regimen), due to overall slow enrollment rate and shifted all relative objectives from primary/secondary to exploratory, due to small sample size.
  Everolimus: in patients randomized to Group A before Amend 1 approval, from the day following randomization, the whole daily dose of everolimus was taken in the morning, at the same time of the CsA and steroid dosing. At the Rand+1W visit, the everolimus dose was adjusted to reach and maintain everolimus blood levels between 5 and 8 ng/mL until end of Month 12.
  Cyclosporine: in patients randomized to Group A before Amend 1 approval, from the day following randomization, the whole cyclosporine daily dose was taken in the morning. The dose was then adjusted to maintain C2 levels between 350 and 700 ng/mL.
  Prednisone: In patients randomized to Group A before Amend 1 approval, the dose of prednisone was kept stable at 5 mg/day in the morning.
- Group B - Steroid Withdrawal Group: Everolimus: after randomization the everolimus dose was adjusted, if necessary, to maintain a C0 within 6-10 ng/mL until M12.
  Cyclosporine: after randomization the cyclosporine dose was adjusted to maintain CsA C2 levels within 300-500 ng/mL until M12.
  Prednisone: starting from Visit 5 (day 90 ± 28 days), oral prednisone was tapered until complete stop. It was recommended to taper prednisone by 1 mg/week until complete stop in 5 to 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Not Randomized Population (NRP) | Group A - Once-a-day Regimen | Group B - Steroid Withdrawal Group | Group C - Standard Twice-a-day Group | Total
Number analyzed (Participants) | 144 | 45 | 68 | 71 | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (11.5) | 46.6 (13.7) | 48.5 (11.6) | 49.2 (13.0) | 50.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 15 | 22 | 20 | 113
  Male | 88 | 30 | 46 | 51 | 215
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 139 | 44 | 68 | 67 | 318
  Black | 3 | 0 | 0 | 1 | 4
  Oriental | 1 | 1 | 0 | 0 | 2
  Other | 1 | 0 | 0 | 3 | 4
Smoking Status [Number; unit: Participants]
  No | 119 | 41 | 58 | 56 | 274
  Yes | 16 | 2 | 2 | 2 | 22
  Missing | 9 | 2 | 8 | 13 | 32
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.6 (3.4) | 24.9 (3.6) | 24.1 (3.3) | 24.2 (3.6) | 24.4 (3.4)
Female reproductive status [Number; unit: Participants]
  Childbearing potential with contraceptive protecti | 11 | 8 | 12 | 4 | 35
  Surgically sterilised | 2 | 0 | 2 | 0 | 4
  Postmenopausal | 43 | 7 | 8 | 16 | 74
Result of HCG pregnancy screen - Negative [Number; unit: Participants]
  Negative | 10 | 6 | 12 | 4 | 32
  Missing | 46 | 9 | 10 | 16 | 81

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure Rate
Description: Occurrence or not of treatment failure in each patient. Treatment failure was defined as a composite endpoint of biopsy-proven acute rejection (a biopsy graded IA, IB, IIA, IIB or III according to Banff '97 grading with 2007 update), graft loss, death or lost to follow-up occurring after randomization (V5) and within M12 (V9).
Time Frame: Between randomization (Month 3) and Month 12
Population: ITT population: all randomized pts who received at least one dose of study drug after Visit 5 & have at least one post-baseline assessment of the primary efficacy variable. Change in study design stopped the randomization into Group A, due to overall slow enrollment rate & shifted all relative objectives to exploratory, due to small sample size.
Measure: Number; unit: Participants
Arm/Group | Group A - Once-a-day Regimen | Group B - Steroid Withdrawal Group | Group C - Standard Twice-a-day Group
Number analyzed (Participants) | 45 | 68 | 71
Participants | 3 | 10 | 2

2. Secondary Outcome: Changes in the Estimated Glomerular Filtration Rate (eGFR) Between Randomization (Month 3) and Month 12
Description: eGFR by Nankivell, in terms of descriptive statistics and change vs randomization visit - to compare the changes in the estimated GFR (Nankivell) between randomization and Month 12 in the steroid withdrawal group (Group B) to the change observed in the standard twice-a-day group (Group C), for non-inferiority
Time Frame: Month 3 to Month 12
Population: ITT population, defined as all randomized patients who received at least one dose of study drug after Visit 5 (Day 90) and have at least one post-baseline assessment of the primary efficacy variable (i.e. treatment failure).
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Group B - Steroid Withdrawal Group | Group C - Standard Twice-a-day Group
Number analyzed (Participants) | 68 | 71
mL/min | -1.7 (9.5) | 2.5 (10.6)

3. Secondary Outcome: Biopsy Proven Acute Rejection (BPAR) Rate Between Randomization and Month 12
Description: Occurrence of BPAR (after randomization) between arm B (steroid withdrawal group) and arm c (standard twice-a-day group).
  BPAR was defined as a biopsy graded IA, IB, IIA, IIB, or III according to Banff 1997 grading with 2007 update.
Time Frame: Month 3 to Month 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Group B - Steroid Withdrawal Group | Group C - Standard Twice-a-day Group
Number analyzed (Participants) | 68 | 71
Participants | 9 | 2

4. Secondary Outcome: Number of Participants With Graft and Patient Survival After Randomization
Description: Graft Survival, calculated from the date of transplantation to the date of irreversible graft failure signified by return to long-term retransplantation or the date of the last follow-up during the period when the transplant was still functioning or to the date of death.
  Patient survival, calculated from the date of transplantation to the date of death or the date of the last follow-up.
Time Frame: Month 3 to Month 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Group B - Steroid Withdrawal Group | Group C - Standard Twice-a-day Group
Number analyzed (Participants) | 68 | 71
Participants | 68 | 71

5. Secondary Outcome: Change in Estimated Creatine Clearance
Description: At each visit, estimated creatinine clearance was measured in the local laboratory to analyze the evolution of the renal function. The following indirect measures of renal function were computed: estimated creatinine clearance according to Cockcroft and Gault formula and MDRD formula.
Time Frame: M3, M12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Group B - Steroid Withdrawal Group | Group C - Standard Twice-a-day Group
Number analyzed (Participants) | 68 | 71
mL/min
  Using Cockcroft and Gault model @ month 3 | 64.8 (21.8) | 63.0 (20.9)
  Using Cockcroft and Gault model @ month 12 | 62.3 (21.4) | 66.9 (24.7)
  Using MDRD-4 formular @ month 3 | 57.9 (20.0) | 58.8 (21.8)
  Using MDRD-4 formular @ month 12 | 53.6 (18.9) | 61.8 (23.1)

6. Secondary Outcome: Change in Serum Creatinine
Description: Serum creatinine (a blood measurement) is an important indicator of renal health because it is an easily-measured by-product of muscle metabolism. Measuring serum creatinine is a simple test and it is the most commonly used indicator of renal function.
Time Frame: M3, M12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group B - Steroid Withdrawal Group | Group C - Standard Twice-a-day Group
Number analyzed (Participants) | 68 | 71
mg/dL
  Serum Creatinine @ month 3 | 1.4 (0.4) | 1.4 (0.4)
  Serum Creatinine @ month 12 | 1.5 (0.5) | 1.4 (0.5)

ADVERSE EVENTS:
Groups:
- Not Randomized Population (NRP): At the Baseline visit, performed up to 48 hours after graft reperfusion, eligible patients entered the Pre-Randomization Period and started study drug treatment (D1 = 1st day of everolimus treatment).
  This population defined in whom a renal transplantation was performed, received at least one dose of study drug (everolimus) but who did not qualify for randomization at Visit 5, Day 90. This group was addressed as "not randomized patients" (NRP) and described with respect to baseline characteristics, treatment and outcome variables.
Arm/Group | Not Randomized Population (NRP) | Group A - Once-a-day Regimen | Group B - Steroid Withdrawal Group | Group C - Standard Twice-a-day Group
Serious Adverse Events (participants affected / at risk) | 65/144 | 18/45 | 24/68 | 25/71
Other Adverse Events (participants affected / at risk) | 108/144 | 35/45 | 56/68 | 57/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Not Randomized Population (NRP) (N=144) | Group A - Once-a-day Regimen (N=45) | Group B - Steroid Withdrawal Group (N=68) | Group C - Standard Twice-a-day Group (N=71)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Device occlusion (General disorders) | 0 | 0 | 1 | 0
Hyperpyrexia (General disorders) | 0 | 0 | 4 | 0
Impaired healing (General disorders) | 1 | 0 | 0 | 0
Implant site haematoma (General disorders) | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 2 | 2 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Kidney transplant rejection (Immune system disorders) | 2 | 2 | 1 | 1
Transplant rejection (Immune system disorders) | 11 | 0 | 6 | 2
Abscess (Infections and infestations) | 0 | 0 | 0 | 1
BK virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 2 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 2
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 1
Human polyomavirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 6 | 0
Wound infection (Infections and infestations) | 2 | 0 | 0 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 4 | 1 | 0 | 0
Graft loss (Injury, poisoning and procedural complications) | 7 | 0 | 0 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 4 | 0 | 3 | 1
Urinary anastomotic leak (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 5 | 2 | 5 | 3
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal artery dissection (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 3 | 0 | 0 | 0
Renal artery thrombosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal cortical necrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 2 | 0
Renal impairment (Renal and urinary disorders) | 5 | 1 | 4 | 6
Renal tubular necrosis (Renal and urinary disorders) | 3 | 0 | 0 | 0
Renal vein thrombosis (Renal and urinary disorders) | 2 | 0 | 0 | 0
Ureteral necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ureteric dilatation (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureteric fistula (Renal and urinary disorders) | 1 | 0 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 1 | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary fistula (Renal and urinary disorders) | 2 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bladder operation (Surgical and medical procedures) | 0 | 0 | 1 | 0
Nephrostomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Ureteral stent removal (Surgical and medical procedures) | 1 | 1 | 0 | 0
Urinary tract operation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Intra-abdominal haematoma (Vascular disorders) | 1 | 0 | 0 | 1
Lymphocele (Vascular disorders) | 2 | 3 | 2 | 1
Lymphorrhoea (Vascular disorders) | 1 | 0 | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Not Randomized Population (NRP) (N=144) | Group A - Once-a-day Regimen (N=45) | Group B - Steroid Withdrawal Group (N=68) | Group C - Standard Twice-a-day Group (N=71)
Anaemia (Blood and lymphatic system disorders) | 53 | 10 | 23 | 13
Leukopenia (Blood and lymphatic system disorders) | 13 | 3 | 5 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 3 | 3 | 1
Atrial fibrillation (Cardiac disorders) | 11 | 1 | 0 | 3
Abdominal hernia (Gastrointestinal disorders) | 0 | 3 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 4 | 1 | 3
Constipation (Gastrointestinal disorders) | 10 | 1 | 1 | 7
Diarrhoea (Gastrointestinal disorders) | 7 | 3 | 8 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 0 | 0
Oedema peripheral (General disorders) | 7 | 6 | 16 | 9
Pyrexia (General disorders) | 14 | 2 | 6 | 2
Urinary tract infection (Infections and infestations) | 25 | 7 | 14 | 16
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 22 | 7 | 6 | 8
Blood creatinine increased (Investigations) | 6 | 6 | 5 | 3
Acidosis (Metabolism and nutrition disorders) | 8 | 0 | 4 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 1 | 2 | 6
Fluid retention (Metabolism and nutrition disorders) | 7 | 2 | 4 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 8 | 3 | 6 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 4 | 4 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 16 | 12 | 20 | 18
Hyperphosphataemia (Metabolism and nutrition disorders) | 8 | 0 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 2 | 3 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 15 | 3 | 7 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 15 | 5 | 7 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 6 | 7 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 6 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 0
Renal impairment (Renal and urinary disorders) | 15 | 3 | 3 | 3
Renal tubular necrosis (Renal and urinary disorders) | 8 | 2 | 3 | 2
Hypertension (Vascular disorders) | 25 | 8 | 11 | 14
Lymphocele (Vascular disorders) | 9 | 5 | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.